CLINICAL TRIAL: NCT02457663
Title: Identification and Validation of Established and Novel Biomarkers for Infections in Burns
Brief Title: Identification and Validation of Biomarkers for Infections in Burns
Status: Terminated | Type: Observational
Why Stopped: At the request of the study site, this study has been closed and access to study-related data is unavailable. We are unable to submit the results-data.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0525
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-02

CONDITIONS: Burns Involving 20% or More of Body Surface
Keywords: Burns
MeSH Terms: conditions — Burns | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood Draw — Blood is to be collected at admission, prior to the 1st operating procedure, once daily for the following 7 consecutive days, at day 15, and at discharge (11 blood draws total). Blood will be taken from IV catheter or routine venipuncture if the catheter is not in place. The blood draw will occur prior to the induction of anesthesia or operating surgical procedure.

SUMMARY:
In this prospective, multi-center study, 200 patients from four participating Texas burn hospitals will be enrolled from admission to discharge. The clinical research study team will collect approximately 11 serum samples and clinical data related to sepsis and infection predictors from severely burned adult patients, ages 18-80 years old. All serum samples from participating sites will be shipped to the lead site, University of Texas Medical Branch. The University of Texas Medical Branch will then validate previously identified biomarkers while simultaneously identifying novel biomarkers through discovery proteomics.

DETAILED DESCRIPTION:
The burn literature is replete with suggested biomarkers of infections for identifying sepsis or other infections in burn patients, however, these reports are largely untested. In order for incorporation of infection biomarker assessment to become the standard of care, validation of these markers in a multi-center prospective study is necessary. As the majority of these biomarkers have been chosen because of success in other patient populations, or ease of measurement, it is possible that the best biomarkers of infection have not yet been discovered in this patient population. Prospective identification and validation of novel biomarkers may also improve early identification of infections in burn patients. Early treatment of infections and sepsis directly correlated with improved survival and reduced costs of care.

In this prospective, multi-center study, 200 patients from four participating Texas burn hospitals will be enrolled from admission to discharge. The clinical research study team will collect approximately 11 serum samples and clinical data related to sepsis and infection predictors from severely burned adult patients, ages 18-80 years old. All serum samples from participating sites will be shipped to the lead site, University of Texas Medical Branch. The University of Texas Medical Branch will then validate previously identified biomarkers while simultaneously identifying novel biomarkers through discovery proteomics.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 years old
* Greater than 20% Total Body Surface Area burn
* Patient arrival to the burn center within 7 days of burn injury

Exclusion Criteria:

* Known history of acquired immunodeficiency syndrome (AIDS), AIDS-related complex (ARC), human immunodeficiency virus (HIV)
* History of cancer within 5 years
* Pregnancy
* Burn injury due to chemical burns or deep electrical injury
* Inability to obtain informed consent
* Decision not to treat due to burn injury severity or futility as deemed by the clinical team at the time of admission (Note: This is a clinical determination of futility beyond which survival is rare. These are typically patients whose sum of Total Body Surface Area % burn and age (Baux score) exceeds 140 or 120 with severe inhalation injury.)
* Presence of anoxic brain injury that is not expected to result in complete recovery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to participating burn centers who meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of infectious and septic episodes | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Celeste C Finnerty, Ph.D., Principal Investigator — University of Texas
Locations (3):
- United States (3):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - U.S. Army Institute of Surgical Research, Fort Sam Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas